CLINICAL TRIAL: NCT02506751
Title: A Phase 1b, Open-label Study to Evaluate the Safety and Tolerability of the Putative Remyelinating Agent, Liothyronine, in Individuals With MS
Brief Title: Open-label Study of Liothyronine in MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061965
Record Dates: First submitted 2015-07-12; First posted 2015-07-23 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liothyronine (Experimental): Subjects will take oral liothyronine for a total of 24 weeks following the below titration schedule:
  0-6 weeks: liothyronine 10mcg po daily (5mcg po BID)
  6-12 weeks: liothyronine 20mcg po daily (10mcg po BID)
  12-18 weeks: liothyronine 50mcg po daily (25mcg po BID)
  18-24 weeks: liothyronine 1mcg/kg/day (0.5mcg/kg po BID), not to exceed 75mcg po daily
  Interventions: Drug: liothyronine

INTERVENTIONS:
Drug: liothyronine — All eligible subjects will be treated with the study drug as per the standardized dose-escalation protocol. Subjects will be required to report to the study site every six weeks for the duration of the study in order to receive their study drug and to monitor drug safety and tolerability.
  Other Names: Cytomel

SUMMARY:
This study will evaluate the safety and tolerability of synthetic T3, liothyronine. It will establish if there are changes in MS symptoms and if there is a positive effect on markers of neuronal health.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, immune-mediated disease of the central nervous system (CNS) that is characterized by inflammation, demyelination, and neurodegeneration. It remains the most common non-traumatic cause of neurologic disability in young adults and presents in most patients as relapsing-remitting disease. Relapses, caused by inflammatory demyelination, can result in a significant amount of neurological disability and reduced health-related quality of life, and having frequent early relapses is associated with increased risk of longer-term disability. Clinical recovery from early relapses is incomplete in approximately half of patients with MS. The mechanisms underlying relapse recovery are not completely understood.

Remyelination of acutely denuded axons is one mechanism by which relapse recovery may occur. Remyelination is suspected to occur via newly differentiated oligodendrocytes, which are derived from oligodendrocyte precursor cells (OPCs) in the CNS. However, despite the presence of this innate repair mechanism, many patients go on to develop progressive functional disability. This may be due to a failure of remyelination or because of progressive axonal injury. Chronic demyelinating lesions are surrounded by OPCs and premyelinating oligodendrocytes, which suggest that failed remyelination does occur and could be partially due to incomplete oligodendrocyte differentiation. Additionally, recent studies have highlighted the importance of mitochondrial dysfunction, perhaps related to oxidative stress or increased energy demands, in mediating MS disease progression. Mitochondrial dysfunction may drive axonal degeneration with resultant neurodegeneration and progressive neurological decline (progressive MS). While numerous immune modulating therapies exist, currently, there is an urgent need for novel therapies that have neuroreparative and neuroprotective properties.

Thyroid hormones may play a direct role in remyelination and repair in the adult CNS by promoting maturation of oligodendrocytes. Further, thyroid hormones have been shown to reduce oxidative stress and thus may have the capacity to prevent mitochondrial dysfunction as well. Since tri-iodothyronine (T3) is believed to mediate the most important thyroid hormone actions, liothyronine (synthetic form of T3) has the potential to induce reparative mechanisms and limit secondary neurodegeneration in MS. In mice, T3 administration has shown to help facilitate recovery from cuprizone-induced demyelination. In this study, the investigators propose to perform a phase 1 study in patients with MS to establish a tolerable dose of liothyronine, evaluate the safety of this medication, determine whether it impacts function, and evaluate if it is associated with changes in neurotrophic and/or inflammatory biomarkers in the cerebrospinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* Must meet 2010 McDonald criteria for clinically definite MS
* Must be euthyroid
* Expanded Disability Status Scale (EDSS) 3.0-7.5
* Patients may be on MS immunomodulating therapies or immunosuppressant therapies during the study

Exclusion Criteria:

* Known thyroid disease (past or current)
* Currently on thyroid replacement therapy
* Steroid use within a month of screening
* History of coronary artery disease, atrial fibrillation, or other clinically significant cardiac disease
* History of adrenal insufficiency
* Ongoing renal and/or liver disease
* Ongoing severe depression and/or anxiety
* Use of carbamazepine, phenytoin, phenobarbital, warfarin, antacids, cholestyramine, colestipol, sucralfate, and rifampin
* Known contraindication to using beta-blocker medications
* History of alcohol or substance abuse in the past 6 months
* Pregnant or nursing
* If the investigator feels that participation in this study is not in the best interest of the subject

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
The incidence rate of adverse events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott Newsome, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Karampampa K, Gustavsson A, Miltenburger C, Eckert B. Treatment experience, burden and unmet needs (TRIBUNE) in MS study: results from five European countries. Mult Scler. 2012 Jun;18(2 Suppl):7-15. doi: 10.1177/1352458512441566. PMID 22623122
- [Background] Orme M, Kerrigan J, Tyas D, Russell N, Nixon R. The effect of disease, functional status, and relapses on the utility of people with multiple sclerosis in the UK. Value Health. 2007 Jan-Feb;10(1):54-60. doi: 10.1111/j.1524-4733.2006.00144.x. PMID 17261116
- [Background] Scott TF, Schramke CJ. Poor recovery after the first two attacks of multiple sclerosis is associated with poor outcome five years later. J Neurol Sci. 2010 May 15;292(1-2):52-6. doi: 10.1016/j.jns.2010.02.008. Epub 2010 Mar 4. PMID 20202650
- [Background] Sormani MP, Li DK, Bruzzi P, Stubinski B, Cornelisse P, Rocak S, De Stefano N. Combined MRI lesions and relapses as a surrogate for disability in multiple sclerosis. Neurology. 2011 Nov 1;77(18):1684-90. doi: 10.1212/WNL.0b013e31823648b9. Epub 2011 Oct 5. PMID 21975200
- [Background] Mowry EM, Pesic M, Grimes B, Deen S, Bacchetti P, Waubant E. Demyelinating events in early multiple sclerosis have inherent severity and recovery. Neurology. 2009 Feb 17;72(7):602-8. doi: 10.1212/01.wnl.0000342458.39625.91. PMID 19221292
- [Background] Chang A, Tourtellotte WW, Rudick R, Trapp BD. Premyelinating oligodendrocytes in chronic lesions of multiple sclerosis. N Engl J Med. 2002 Jan 17;346(3):165-73. doi: 10.1056/NEJMoa010994. PMID 11796850
- [Background] Witte ME, Bo L, Rodenburg RJ, Belien JA, Musters R, Hazes T, Wintjes LT, Smeitink JA, Geurts JJ, De Vries HE, van der Valk P, van Horssen J. Enhanced number and activity of mitochondria in multiple sclerosis lesions. J Pathol. 2009 Oct;219(2):193-204. doi: 10.1002/path.2582. PMID 19591199
- [Background] van Horssen J, Witte ME, Ciccarelli O. The role of mitochondria in axonal degeneration and tissue repair in MS. Mult Scler. 2012 Aug;18(8):1058-67. doi: 10.1177/1352458512452924. Epub 2012 Jun 21. PMID 22723572
- [Background] Harsan LA, Steibel J, Zaremba A, Agin A, Sapin R, Poulet P, Guignard B, Parizel N, Grucker D, Boehm N, Miller RH, Ghandour MS. Recovery from chronic demyelination by thyroid hormone therapy: myelinogenesis induction and assessment by diffusion tensor magnetic resonance imaging. J Neurosci. 2008 Dec 24;28(52):14189-201. doi: 10.1523/JNEUROSCI.4453-08.2008. PMID 19109501